CLINICAL TRIAL: NCT02468401
Title: The Efficacy of a New Protocol for Preventing Contrast Induced Nephropathy in Patients With Advanced Renal Dysfunction Undergoing Coronary Interventions
Brief Title: Prevention of Contrast Induced Nephropathy in Patients With Advanced Renal Dysfunction Undergoing Coronary Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Pereg David, Dr, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0103-15-MMC
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Disease, Chronic; Ischemic Heart Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

ARMS (1):
- Coronary angiography (Experimental): Patients undergoing coronary angio with or without percutaneous coronary intervention using a new protocol designed to minimize the exposure to contrast medium
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Patients planned for coronary angiography or percutaneous coronary intervention will be managed using a protocol that allows us to use minimal volumes of contrast dye

SUMMARY:
There is a pressing need to find effective strategies for the prevention of contrast induced nephropathy in patients with advanced renal dysfunction. The current study was designed to assess the efficacy of a new protocol for preventing contrast induced nephropathy in patients with advanced renal dysfunction undergoing coronary interventions

ELIGIBILITY:
Inclusion Criteria:

Patients with estimated glomerular filtration rate<45ml/min undergoing coronary angiography due to one of the following indications in accordance with the 2014 guidelines:

1. Elective coronary angiography due to symptoms suggestive for angina with a positive non-invasive ischemia assessment of ≥10% of left ventricle.
2. Non ST-elevation acute coronary syndrome with a GRACE score>110

Exclusion Criteria:

* Patients on dialysis or those planned for dialysis in the next 3 months.
* Patients with ST-elevation myocardial infarction
* No symptoms or signs of heart failure
* Treatment with IV diuretics during the 48 hours prior to enrolment
* Patients with acute renal failure (Creatinine raise of at least 0.3mg/dl from )baseline
* Patients post coronary artery bypass surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes in glomerular filtration rate following coronary angiography or intervention | 24 and 48 hours post procedure
  Significant changes are defined as a reduction ≥25% in glomerular filtration rate

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel

REFERENCES:
- [Derived] Rozenbaum Z, Benchetrit S, Rozenbaum E, Neumark E, Mosseri M, Pereg D. Ultra-Low Contrast Volume for Patients with Advanced Chronic Kidney Disease Undergoing Coronary Procedures. Nephron. 2018;138(4):296-302. doi: 10.1159/000485648. Epub 2018 Jan 24. PMID 29393219